CLINICAL TRIAL: NCT04342273
Title: A Through QT/QTc Study of KW-6356 in Japanese Healthy Adults
Brief Title: A Through QT/QTc Study of KW-6356
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6356-007
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KW-6356 therapeutic dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- KW-6356 supratherapeutic dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- Placebo (Placebo Comparator): Oral administration
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Oral administration
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: KW-6356 — KW-6356 will be administered once daily as therapeutic at Day 1 through Day 7
  Arms: KW-6356 therapeutic dose
Drug: KW-6356 — KW-6356 will be administered once daily as supratherapeutic dose at Day 1 through Day 7
  Arms: KW-6356 supratherapeutic dose
Drug: Placebo — Placebo will be administered once daily at Day 1 through Day 7
  Arms: Placebo
Drug: Moxifloxacin — Placebo will be administered once daily at Day 1 through Day 6, followed by Moxifloxacin once daily at Day 7.
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the effects of multiple therapeutic and supratherapeutic doses of KW-6356 on the QT interval corrected for heart rate in Japanese healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having issued written consent to this study at their own discretion
* Men or women aged 20 to 54 years at the time of informed consent
* Subjects with BMI ≥18.5 and <25.0 at screening
* In case of women of childbearing potential,* subjects who have agreed to use highly effective and appropriate contraceptive methods from the time of informed consent to 4 weeks after the last dose of the investigational product or the index drug. Women of childbearing potential must have a negative serum pregnancy test at screening
* At screening and Day -2, subjects with resting pulse rate of ≥45 and <100 bpm, systolic blood pressure of ≥90 and <140 mmHg, and diastolic blood pressure of ≥40 and <90 mmHg when measured in the supine position
* Subjects whose standard 12-lead ECG data obtained at screening and Day -2 meet the following criteria and show no clinically significant abnormalities as confirmed by the investigator or subinvestigator Normal sinus rhythm: HR of ≥45 and ≤100 bpm QTc interval (QTcF): ≤450 msec QRS interval: ≤120 msec (must be re-measured manually if exceeding 120 msec) PR interval: ≤220 msec
* Subjects whose potassium, sodium, calcium, and magnesium levels at screening are within institutional normal limits

Exclusion Criteria:

* Subjects with any current disease requiring treatment
* Subjects having drug allergy or its history
* Subjects having psychiatric disease or its history
* Positive results for any of the following infection-related items examined at screening: hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, human T-lymphotropic virus (HTLV)-1 antibody, rapid plasma reagin (RPR) test, or Treponema pallidum (TP) antibody
* Subjects being alcohol- or drug-dependent or having a positive result for any of the drug abuse test items
* Subjects previously or concurrently having any of the following diseases or subjects with a family history of any of the following diseases:

Hypokalemia, hypocalcemia, and/or long QT syndrome Risk factors for torsade de pointes such as cardiac failure, cardiomyopathy, and a family history of long QT syndrome Sick sinus syndrome, second- or third-degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, QT interval prolongation, or atrioventricular conduction disturbance Repeated or frequent syncope or vasovagal attack Hypertension, angina pectoris, bradycardia, or severe peripheral arterial circulatory disorder

* Subjects categorized as patients listed in the warnings or contraindications section of the package insert of moxifloxacin hydrochloride
* Subjects unable to be compliant with Specified "Concomitant Medication and Concomitant Therapy" and "Instruction for Subjects"
* Subjects having participated in a clinical study of a pharmaceutical product or a medical device or any equivalent study and used the investigational product or the unapproved medical device within 4 months prior to administration of the investigational product
* Subjects having used any drug within 2 weeks prior to administration of the investigational product
* Subjects having consumed grapefruit or any food or beverage containing St John's wort within 1 week prior to administration of the investigational product
* Subjects having smoked or used smoking cessation agents within 4 weeks prior to administration of the investigational product
* Subjects categorized as "yes" to "active suicidal ideation with some intent to act, without specific plan" or "active suicidal ideation with specific plan and intent" on the Columbia-Suicide Severity Rating Scale assessed on Day -2 or subjects with a history of or currently observed suicidal behavior
* Subjects having undergone ≥400 mL of blood collection within 12 weeks prior to administration of the investigational product or ≥200 mL of blood collection within 4 weeks prior to administration of the investigational product for blood donation or in a clinical trial, etc. or subjects having undergone blood collection for pheresis donation within 2 weeks prior to administration of the investigational product
* Subjects having issued no consent to adoption of any appropriate contraceptive method during the period from day of informed consent to 4 weeks after the final administration of the investigational product or the index drug for women of childbearing potential and during the period from start day of study treatment to 12 weeks after the final administration of the investigational product or the index drug for men of reproductive potential. The appropriate contraceptive method

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTc interval [QTcF] (ΔQTcF) | Day 1 through Day 7

SECONDARY OUTCOMES:
Changes from baseline in the HR | Day 1 through Day 7
Changes from baseline in the QTc interval [QTcF] | Day 1 through Day 7
Changes from baseline in the PR interval | Day 1 through Day 7
Changes from baseline in the QRS interval | Day 1 through Day 7
Placebo-corrected ΔQTcF | Day 1 through Day 7
Placebo-corrected ΔHR | Day 1 through Day 7
Placebo-corrected ΔPR interval | Day 1 through Day 7
Placebo-corrected ΔQRS interval | Day 1 through Day 7
Outliers in terms of category for HR | Day 1 through Day 7
Outliers in terms of category for QTc interval (QTcF) | Day 1 through Day 7
Outliers in terms of category for PR interval | Day 1 through Day 7
Outliers in terms of category for QRS interval | Day 1 through Day 7
Frequency of morphological changes in T wave after administration of the investigational product | Day 1 through Day 7
Frequency of morphological changes in U wave after administration of the investigational product | Day 1 through Day 7
Incidence of treatment-emergent adverse events | Day 1 through Day 20
Plasma concentrations of KW-6356 | Day 1 through Day 8, and Day 12

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Medical Co. LTA Sumida Hospital, Sumida-ku, Tokyo
  - Medical Co. LTA Fukuoka Mirai Hospital Clinical Research Center, Fukuoka

IPD SHARING:
Plan to Share IPD: Undecided